CLINICAL TRIAL: NCT00220727
Title: Randomized, Controlled, Open Study Investigating IGIV-C, 10% Given at Different Infusion Rates on Intravascular Hemolysis in Patients With Idiopathic (Immune) Thrombocytopenic Purpura (ITP)
Brief Title: Rapid Infusion Of Immune Globulin Intravenous (IGIV) In Patients With ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 100422
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: Idiopathic (Immune) Thrombocytopenic Purpura; Immunoglobulin G
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombocytopenic | interventions — gamma-Globulins; Caprylates; Immunoglobulins, Intravenous; Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Infusion #1 (Week 0) IGIV-C (0.08 mL/kg/min); Infusion #2 (Week <6) IGIV-C (0.14 mL/kg/min)
  Interventions: Drug: Immune Globulin IV [Human], 10% Caprylate/Chromatography Purified
- Group 2 (Experimental): Infusion #1 (Week 0) IGIV-C (0.14 mL/kg/min); Infusion #2 (Week <6) IGIV-C (0.08 mL/kg/min)
  Interventions: Drug: Immune Globulin IV [Human], 10% Caprylate/Chromatography Purified

INTERVENTIONS:
Drug: Immune Globulin IV [Human], 10% Caprylate/Chromatography Purified — IGIV-C 10% at a dose of 1.0g/kg was to be given on 2 occasions as a single daily infusion: Group 1 were to receive their first IGIV-C, 10-% infusion at a rate of 0.08 mL/kg/min and a second infusion at 0.14 mL/kg/min. and Group 2 were to receive their first IGIV-C, 10-% infusion at a rate of 0.14 mL/kg/min and a second infusion at a rate of 0.08 mL/kg/min.
  Other Names: Gamunex®; IGIVnex®; Gaminex; IGIV-C; IGIV-C, 10%; IVIG; BAY 41-1000; TAL-05-00004; Immune Globulin (Human), 10% (IGIV); Immune Globulin Intravenous, 10% by Chromatography Process; NDC 13533-645-12; NDC 13533-645-15; NDC 13533-645-20; NDC 13533-645-24; NDC 13533-645-71

SUMMARY:
The objective of this study is to determine if the safety and tolerability of Immune Globulin Intravenous (Human), 10% Caprylate/Chromatograph Purified (IGIV-C) is similar when infused at two different infusion rates.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center, open, cross-over trial in patients with a confirmed diagnosis of Idiopathic Thrombocytopenia Purpura (ITP). ITP is defined as isolated thrombocytopenia in a patient with no other clinically apparent associated conditions or factors that are known to cause thrombocytopenia as defined by the ITP Practice Guidelines Committee of the American Society of Hematology.

Immune Globulin Intravenous (Human), 10% Caprylate/Chromatography Purified (IGIV-C) at a dose of 1.0 g/kg will be given on 2 occasions as a single daily infusion for platelet counts < 30,000 microliters (uL) or if clinically indicated, at maximum intervals of six weeks. Eligible patients will be randomized into one of two cross-over groups. Patients randomized to Group 1 will receive their first IGIV-C infusion at a rate of 0.08 mL/kg/min and their second infusion at a rate of 0.14 mL/kg/min. Conversely patients randomized to Group 2 will receive their first IGIV-C infusion at a rate of 0.14 mL/kg/min and their second infusion at a rate of 0.08 mL/kg/min according to the following schema:

Group 1:

* Infusion #1 (Week 0) IGIV-C (0.08 mL/kg/min)
* Infusion #2 (Week <6) IGIV-C (0.14 mL/kg/min)

Group 2:

* Infusion #1 (Week 0) IGIV-C (0.14 mL/kg/min)
* Infusion #2 (Week <6) IGIV-C (0.08 mL/kg/min)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from patient or legal guardian (according to institutional review board requirements)obtained prior to initiation of any study related procedures
* Male and female subjects age between 12 and 75 years
* Confirmed diagnosis of ITP logged in medical records available prior to entry into the trial.
* Patients must have a platelet count < 30 x Giga/L (this level can be higher if clinically indicated).
* Previously splenectomized patients may be included.
* Any previously conducted bone marrow aspirations if conducted following diagnosis of ITP must be consistent with the ITP diagnosis (increased or normal levels of megakaryocytes in otherwise normal bone marrow).

Exclusion Criteria:

* History of allergic or other clinically significant reaction to human gamma globulin or other plasma proteins and/or blood products.
* Female patient who is pregnant or lactating or is not on an adequate program of contraception if of child-bearing potential.
* Documented history of selective immunoglobulin A (IgA) deficiency (serum <5.0 mg/dL) and known antibodies to IgA.
* Currently on intermittent prednisone therapy. Prednisone therapy is allowed only if the patient has been on stable daily doses of prednisone for the preceding month and maintains the same treatment regimen throughout the study.
* Renal or liver impairment defined by creatinine > 2.5 mg/dL, or direct bilirubin >1.5 X the upper limit of normal or liver transaminases (AST or ALT) > 3 times the upper limit of normal.
* Received anti-D or IGIV infusions within the past 14 days
* Pre-treatment with the exception of acetominophen, routinely required to control/ameliorate IGIV infusion-related adverse events (AEs), or any patient who has been, unresponsive to IGIV therapy for their ITP
* History or clinical evidence of medical conditions felt to be the underlying cause of their thrombocytopenia. Such conditions commonly include systemic lupus erythematosus, history of chronic lymphocytic leukemia, dysplasia, agammaglobulinemia, treatment with heparin, quinidine, quinine, trimethoprim-sulfamethoxazole, or ticlopidine or any other drug thought to be the cause of patient's thrombocytopenia, congenital or hereditary thrombocytopenia, or pseudothrombocytopenia (clumping on peripheral blood smear)
* Conditions that could alter protein catabolism and/or immunoglobulin G (IgG) utilization (e.g. protein-losing enteropathies, nephrotic syndrome)
* Congestive heart failure (New York Heart Association Stage III or IV)
* Diabetes mellitus
* Paraproteinemia
* Concomitant nephrotoxic drugs
* Hemoglobin level more than 2g/L below the lower limit of normal.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-07; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Bussel, MD, Principal Investigator — New York Presbyterian Hospital-Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Background] Bussel JB, Hanna K; IGIV-C in ITP Study Group. Safety and tolerability of a novel chromatography-based intravenous immunoglobulin when administered at a high infusion rate in patients with immune thrombocytopenic purpura. Am J Hematol. 2007 Mar;82(3):192-8. doi: 10.1002/ajh.20822. PMID 17109385
- See also: FDA-Approved Product Labeling - Gamunex® — http://www.talecris-pi.info/inserts/gamunex.pdf
- See also: FDA Product Approval - Gamunex® — http://www.fda.gov/BiologicsBloodVaccines/BloodBloodProducts/ApprovedProducts/LicensedProductsBLAs/FractionatedPlasmaProducts/ucm089390.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single-center, open label study in patients with a confirmed diagnosis of Idiopathic Thrombocytopenic Purpura (ITP).
Groups:
- IGIV-C, 10% - 0.08/0.14 mL/kg/Min: Infusion #1 (Week 0 IGIV-C (0.08 mL/kg/min); Infusion #2 (Week <6) IGIV-C (0.14 mL/kg/min)
- IGIV-C, 10% - 0.14/0.08 mL/kg/Min: Infusion #1 (Week 0) IGIV-C (0.14 mL/kg/min); Infusion #2 (Week <6) IGIV-C (0.08 mL/kg/min)
Period: First Infusion (Week 0)
Arm/Group | IGIV-C, 10% - 0.08/0.14 mL/kg/Min | IGIV-C, 10% - 0.14/0.08 mL/kg/Min
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Second Infusion (Week <6)
Arm/Group | IGIV-C, 10% - 0.08/0.14 mL/kg/Min | IGIV-C, 10% - 0.14/0.08 mL/kg/Min
Started | 4 | 4
Completed | 3 | 4
Not Completed | 1 | 0
Not completed — Pt did not meet study requirement | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGIV-C, 10% - 0.08/0.14 mL/kg/Min | IGIV-C, 10% - 0.14/0.08 mL/kg/Min | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.75 (15.78) | 47.50 (14.89) | 47.63 (14.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Free Hemoglobin
Description: Free hemoglobin as a measure to assess hemolysis.
Time Frame: 24 hours after treatment
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- IGIV-C, 10% (0.08 mL/kg/Min): Infusion #1 (Week 0 IGIV-C (0.08 mL/kg/min); Infusion #2 (Week <6) IGIV-C (0.14 mL/kg/min)
- IGIV-C, 10% (0.14 mL/kg/Min): Infusion #1 (Week 0) IGIV-C (0.14 mL/kg/min); Infusion #2 (Week <6) IGIV-C (0.08 mL/kg/min)
Arm/Group | IGIV-C, 10% (0.08 mL/kg/Min) | IGIV-C, 10% (0.14 mL/kg/Min)
Number analyzed (Participants) | 7 | 7
g/dL | 13.057 (1.778) | 12.371 (2.644)

2. Secondary Outcome: Number of Subjects With Infusion Related Adverse Events
Time Frame: 48 hours after treatment
Measure: Number; unit: participants
Groups:
- IGIV-C, 10% (0.08 mL/kg/Min): Slow Infusion Rate IGIV-C (0.08 mL/kg/min);
- IGIV-C, 10% (0.14 mL/kg/Min): Rapid Infusion Rate IGIV-C (0.14 mL/kg/min);
Arm/Group | IGIV-C, 10% (0.08 mL/kg/Min) | IGIV-C, 10% (0.14 mL/kg/Min)
Number analyzed (Participants) | 3 | 4
participants | 2 | 3

3. Primary Outcome: Hematocrit
Description: Hematocrit as a measure to assess hemolysis
Time Frame: 24 hrs after treatment
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | IGIV-C, 10% (0.08 mL/kg/Min) | IGIV-C, 10% (0.14 mL/kg/Min)
Number analyzed (Participants) | 7 | 7
percentage of blood | 36.80 (4.711) | 35.043 (6.793)

4. Primary Outcome: Red Blood Cells
Description: Red blood cells as a measure to assess hemolysis
Time Frame: 24 hrs after treatment
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | IGIV-C, 10% (0.08 mL/kg/Min) | IGIV-C, 10% (0.14 mL/kg/Min)
Number analyzed (Participants) | 7 | 7
10^12 cells/L | 4.1514 (.4820) | 4.0786 (0.8258)

5. Primary Outcome: Change From Baseline in Platelet Levels
Time Frame: 24 hours Post infusion and Day 7
Measure: Mean (Standard Deviation); unit: Giga/L
Arm/Group | IGIV-C, 10% (0.08 mL/kg/Min) | IGIV-C, 10% (0.14 mL/kg/Min)
Number analyzed (Participants) | 6 | 7
Giga/L
  Baseline | 29.50 (28.47) | 6.86 (3.39)
  24 hours post infusion | 21.17 (35.49) | 42.29 (12.41)
  Day 7 | 76 (138.35) | 118.7 (165.80)

ADVERSE EVENTS:
Groups:
- IGIV-C, 10% - 0.08 mL/kg/Min: IGIV-C (0.08 mL/kg/min);
- IGIV-C, 10% - 0.14 mL/kg/Min: IGIV-C (0.14 mL/kg/min);
Arm/Group | IGIV-C, 10% - 0.08 mL/kg/Min | IGIV-C, 10% - 0.14 mL/kg/Min
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGIV-C, 10% - 0.08 mL/kg/Min (N=8) | IGIV-C, 10% - 0.14 mL/kg/Min (N=7)
Abdominal Distention (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will be free to disclose at scientific meetings and to publish in the scientific literature data resulting from these trials. A copy of any manuscript must be sent to sponsor for review at least 1 month prior to submission for publication.